CLINICAL TRIAL: NCT02342145
Title: Efficacy of Basiliximab in the Prevention of Acute Graft-versus-host Disease in Unrelated Allogeneic Hematopoietic Stem Cell Transplantation Therapy for Thalassemia Major Treatment: a Multi-center, Open, Randomized, Controlled Clinical Study
Brief Title: Efficacy of Basiliximab in the Prevention of Acute Graft-versus-host Disease in Unrelated Allogeneic Hematopoietic Stem Cell Transplantation Therapy for Thalassemia Major
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhongming Zhang (Other)
Collaborators: Liuzhou Workers' Hospital (Other Government); Hainan General Hospital (Other); McMaster University (Other); Guangxi Key Laboratory of Thalassemia Research (Unknown); NHC Key Laboratory of Thalassemia Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Zhongming Zhang, The First Affiliated Hospital of Guangxi Medical University, First Affiliated Hospital of Guangxi Medical University
Organization: First Affiliated Hospital of Guangxi Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: gxmuh-2014-14
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Beta-Thalassemia Major; Graft-versus-host Disease (GVHD)
Keywords: beta-Thalassemia major; Graft-versus-host disease; Basiliximab; Allogeneic hematopoietic stem cell transplantation; matched unrelated donors
MeSH Terms: conditions — beta-Thalassemia; Graft vs Host Disease | interventions — Basiliximab; Tacrolimus; Methotrexate; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group A (Experimental): The patients were used FK506 (0.03mg/kg/day), Methotrexate (15mg/m2 on +1d, 10mg/m2 on +3d, +6d, +11d), Mycophenolate Mofetil (0.25g/d, days-1 to 90) and Basiliximab (use 10mg for weight under 35kg, 20mg for over 35kg, 0d and +4d) for prevention of acute graft-versus-host-disease.
  Interventions: Drug: Basiliximab,; Drug: Tacrolimus; Drug: Methotrexate; Drug: Mycophenolate mofetil
- group B (Active Comparator): The patients were used FK506 (0.03mg/kg/day), Methotrexate (15mg/m2 on +1d, 10mg/m2 on +3d, +6d, +11d), Mycophenolate Mofetil (0.25g/d, days-1 to 90) for prevention of acute graft-versus-host-disease.
  Interventions: Drug: Tacrolimus; Drug: Methotrexate; Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Basiliximab, — Basiliximab was used on 0d (after transplantation) and +4d (10mg for weight under 35kg, 20mg for over 35kg) .
  Other Names: chimeric mouse-human antiCD25
  Arms: group A
Drug: Tacrolimus — Specifically Tacrolimus was used by intravenous drip infusion on 0.03mg/kg dosage from -1d and change to 0.1mg/kg oral when gastrointestinal function recovers. The blood concentrations of cyclosporine A was maintained 5-10 ng/ml.
  Other Names: FK506
Drug: Methotrexate — Methotrexate was used 15mg/m2 on +1d and 10mg/m2 on +3d,+6d,+11d by intravenous for prevention of graft-versus-host-disease.
  Other Names: Ametnopterin
Drug: Mycophenolate mofetil — Mycophenolate mofetil was used 0.25g per day from -1d to 90d for prevention of graft-versus-host-disease.
  Other Names: Mycophenolic acid

SUMMARY:
The purpose of this study is to evaluate the basiliximab for prevention of graft-versus-host disease in unrelated allo-genetic hematopoietic stem cell transplantation for thalassemia major. The objective was to evaluate the effect and safety of basiliximab for acute graft-versus-host disease.

DETAILED DESCRIPTION:
Allo-geneic stem cell transplantation(allo-HSCT) cure thalassemia major by destroying the original hematopoietic and immune systems with a large dose of chemotherapy, rebuilding a new system to correct the abnormal hematopoietic globin chain synthesis which leads to hemolysis. Currently, it is the only curative means. According to donors, allo-HSCT could be sibling allogeneic hematopoietic stem cell transplantation and unrelated allogeneic hematopoietic stem cell transplantation(URD-HSCT). URD-HSCT could expand the range of treatment among β-thalassemia major patients. As recently reported , 68 cases of thalassemia patients at the median age of 15 (2 to 37 ) received unrelated donor BMT. According to Pesaro rating classification, 14 patients were attributed to type Ⅰ, 16 cases Ⅱ type , 38 cases type III, overall survival and thalassemia free survival rates were 79.3% and 65.8%. A survey among 59 evaluable patients indicated that grade Ⅱ ~ Ⅳ aGVHD occurred in 24 cases (40%) , in which 10 cases (17%) were grade Ⅲ ~ Ⅳ aGVHD. Similar results were seen in other reports, 21 patients received unrelated donor BMT, with a 2-year thalassemia free survival rate of 71%. GVHD happened in 3 cases, and 3 patients died. Our institution has conducted a total of 10 cases of URD-HSCT to treat severe thalassemia, using methotrexate + cyclosporine A+ mycophenolate mofetil to prevent graft-versus-host disease, 9 cases of disease-free survival, 1 case with graft rejection. Incidence of Ⅲ-Ⅳ severe acute graft-versus-host disease (aGVHD) was 20%. Severe aGVHD incidence was 20%. Our research group has found there is a high risk to develop aGVHD, especially severe aGVHD for heavy thalassemia patients who receive URD-HSCT, which seriously affects the prognosis and survival, while increasing medical costs and the financial burden on the patients' families.

The key factor affecting URD-HSCT's success is GVHD. Thus effective prevention and treatment of GVHD is a prerequisite to ensure a successful transplant. CD25 is a humanized monoclonal IgG1,with murine anti-human IL-2RA chain complement determining region retained. IL-2RA chain expressed only on the surface of activated cytotoxic T cells, which could convert the IL-2R complexes into a higher affinity. The feature that IL-2RA distributes only on the surface of activated lymphocytes indicates it's a ideal target when designing the policy to scavenge antigen-specific allogeneic reactive T cells. In vitro experiments, CD25 monoclonal antibody binds specifically with IL-2RA+ cells by inhibiting IL-2 binding to its receptor competitively. Basiliximab has now been used as first-line medication for aGVHD treatment, as well as the combined prevention of hematologic malignancies URD-HSCT treatment . However as for thalassemia major URD-HSCT, few cases have been reported.

This study was aimed at the high incidence of aGVHD, especially severe aGVHD in thalassemia major URD-HSCT. Basiliximab was added to the original prevention program. The aGVHD incidence, implantation rate, transplant-related mortality, infection incidence would be observed. It is hopeful to reduce the aGVHD incidence after URD-HSCT and promote curative effect.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of TM with hemoglobin electrophoresis, a genetic diagnosis of -thalassemia by DNA analysis, and blood transfusion dependence;
2. a cardiac ejection fraction >50%;
3. normal pulmonary function tests and pulmonary examination results;
4. normal kidney function.

Exclusion Criteria:

1. aspartate aminotransferase level >4- fold the upper limit of normal range in our institution's laboratory criteria;
2. uncontrolled bacterial, viral, or fungal infection;
3. positive serology for HIV;
4. cytomegalovirus (CMV) or Epstein-Barr virus (EBV) copy number >200 copies/mL in blood by quantitative PCR. Patients positive for hepatitis C or hepatitis B virus were also excluded.

(8) Other circumstances which do not meet the inclusion criteria

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
grade II-IV acute graft-versus-host disease incidence | 100 days after matched unrelated donor hematopoietic stem cell transplantation.
  The cumulative incidence of grade II-IV acute graft-versus-host disease after matched unrelated donor hematopoietic stem cell transplantation +100d.

SECONDARY OUTCOMES:
Implantation rate | three years
Transplanted-related mortality | three years
Infection incidence | three years
  CMV reactivation, EBV reactivation, bacterial infection, fungal infection, etc.
Chronic graft-versus-host-disease incidence | five years
Overall survival | three years
Disease-free-survival | three years

CONTACTS AND LOCATIONS:
Overall Officials: yongrong lai, PhD, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (3):
- China (3):
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - The affiliated hospital of guangxi medical university, Nanning, Guangxi
  - Hainan general Hospital, Haikou, Hainan

REFERENCES:
- [Background] Smiers FJ, Krishnamurti L, Lucarelli G. Hematopoietic stem cell transplantation for hemoglobinopathies: current practice and emerging trends. Pediatr Clin North Am. 2010 Feb;57(1):181-205. doi: 10.1016/j.pcl.2010.01.003. PMID 20307718
- [Background] Feng Z, Sun E, Lan H, Zhang C, Li Q, Zhu W. Unrelated donor bone marrow transplantation for beta-thalassemia major: an experience from China. Bone Marrow Transplant. 2006 Jan;37(2):171-4. doi: 10.1038/sj.bmt.1705193. PMID 16273116
- [Background] Hongeng S, Pakakasama S, Chuansumrit A, Sirachainan N, Kitpoka P, Udomsubpayakul U, Ungkanont A, Jootar S. Outcomes of transplantation with related- and unrelated-donor stem cells in children with severe thalassemia. Biol Blood Marrow Transplant. 2006 Jun;12(6):683-7. doi: 10.1016/j.bbmt.2006.02.008. PMID 16737942
- [Background] Wang HX, Yan HM, Wang ZD, Xue M, Liu J, Guo ZK. Haploidentical hematopoietic stem cell transplantation in hematologic malignancies with G-CSF mobilized bone marrow plus peripheral blood stem cells grafts without T cell depletion: a single center report of 29 cases. Leuk Lymphoma. 2012 Apr;53(4):654-9. doi: 10.3109/10428194.2011.624225. Epub 2011 Dec 5. PMID 21929286
- [Background] Hu LD, Chen H, Jiang M, Li BT, Yu ZY, Li YH. [The role of CD25 antibody in unrelated hematopoietic stem cell transplantation]. Zhonghua Nei Ke Za Zhi. 2005 Nov;44(11):848-50. Chinese. PMID 16316569